CLINICAL TRIAL: NCT04224935
Title: The Effect of Leukocyte Platelet Rich Fibrin(L-PRF) Membrane in The Treatment of Localized Gingival Recession (Randomized Controlled Clinical Trial)
Brief Title: The Effect of (L-PRF) Membrane in The Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Zainab Hafez Abdel Rahman, teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 453
Record Dates: First submitted 2020-01-01; First posted 2020-01-13 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Localized Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leukocyte Platelet Rich Fibrin (Active Comparator): Leukocyte Platelet Rich Fibrin will be used
  Interventions: Procedure: Leukocyte Platelet rich fibrin membrane
- connective tissue (Active Comparator): connective tissue will be used
  Interventions: Procedure: Leukocyte Platelet rich fibrin membrane

INTERVENTIONS:
Procedure: Leukocyte Platelet rich fibrin membrane — the use of Leukocyte Platelet rich fibrin as grafting materials for treatment of recession
  Other Names: sub epithelial connective tissue

SUMMARY:
evaluation of the use of L-PRF membrane with coronally repositioned flap in treatment of localized gingival recession (Class I & II) in comparison with the use of connective tissue graft

DETAILED DESCRIPTION:
Twenty patients, who are candidates for gingival recession coverage, will participate in this prospective clinical trial.

Group 1(10 patients) :

Coronally repositioned flap will be done and L PRF membrane will be placed into the tissues

Group 2 (Control group)(10 patients) :

Coronally repositioned flap will be done with sub epithelial connective tissue Parameters

* Clinical evaluation of percentage of root coverage and keratinized tissue width
* Esthetic outcome evaluation Will be done using the root coverage esthetic score (Cairo et al. 2009) that include

Both evaluations will be done at 3, 6 and 9 months

ELIGIBILITY:
Inclusion Criteria:

* Systemically free patients (American Society of Anesthesiologists I; ASA I).
* Age range (20 -40) years.
* Good compliance with the plaque control instructions following initial therapy.
* Patients diagnosed with Miller class I or II in anterior and premolar teeth
* Availability for follow up and maintenance program.

Exclusion Criteria:

* Patient suffering from periodontitis
* Presence of smoking habit.
* Presence of occlusion interference.
* Pregnant and lactating females.
* Vulnerable group of patients (handicapped, mentally retarded and prisoners).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
recession treatment | 9 months
  2-Esthetic outcome evaluation was done using Root coverage esthetic score (RES) system ( Cairo et al. 2009) the RES include the following parameters
  • Level of the gingival margin (GM):(minimum) Zero points = failure of root coverage (gingival margin apical or equal to the baseline recession); 3 points = partial root coverage;(maximum) 6 points = CRC.

SECONDARY OUTCOMES:
soft tissue thickness (Volumetric assessment) | 9 months
  Preoperatively a cast was made and scanned. At 9 months after surgical procedure the same procedure was done to determine the soft tissue thickness after the surgery. The difference between the tissue thickness before and after was used to determine the efficacy of the different surgical grafting materials used.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abdel aziz, co professor, Study Chair — faculty of dentistry ain shams university
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT04224935/Prot_001.pdf